CLINICAL TRIAL: NCT05053230
Title: Integrative Medicine for Patient-reported Outcomes, Values, and Experience (IMPROVE)
Brief Title: A Study Evaluating the Integrative Medicine at Home (IM@HOME) Program in People With Cancer
Acronym: IMPROVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-369
Record Dates: First submitted 2021-09-20; First posted 2021-09-22 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Head and Neck Cancer; Head and Neck Tumor; Thoracic Tumor; Thoracic Cancer; Gynecologic Cancer; Gynecologic Tumor; Melanoma; Ovarian Cancer
Keywords: Head and Neck Cancer; head and neck tumor; thoracic tumors; gynecological tumors; melanoma; 21-369; Memorial Sloan Kettering Cancer Center; ovarian cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Thoracic Neoplasms; Genital Neoplasms, Female; Melanoma; Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IM@Home (Experimental): Participants with head and neck tumors, thoracic tumors, gynecological tumors, melanoma, breast cancer, or ovarian cancer
  Interventions: Behavioral: IM@Home
- Enhanced usual care (Other): Participants with head and neck tumors, thoracic tumors, gynecological tumors, melanoma, breast cancer, or ovarian cancer
  Interventions: Behavioral: Enhanced usual care

INTERVENTIONS:
Behavioral: IM@Home — Participants in the IM@Home group will receive a 12-week virtual, synchronous, mind-body and fitness program. The Classes will be conducted via Zoom video conferencing platform. Patients will choose from a variety of weekly classes, occurring one to four times per week. An Integrative Medicine Service (IMS) clinical therapist (e.g., licensed dance therapist, certified yoga instructor, nurse specialist/physical trainer) with specific expertise in the oncology setting will lead each session. Activities range from more movement-based (fitness, yoga, dance therapy, or tai chi) to meditative-based classes (meditation, guided meditation, or music therapy). All clinicians will provide an overview of the session, 25 to 40 minutes of content, and five minutes for feedback and discussion. Each class lasts 30 to 45 minutes with optional audio or video participant participation and group chat.
  Arms: IM@Home
Behavioral: Enhanced usual care — Patients in the enhanced usual care will receive usual care. In addition, once enrolling into the trial, they will be given a handout to encourage them to visit the MSK's multimedia page on the Integrative Medicine website to access pre-recorded, on-demand meditation audio or video recordings for meditation, guided imagery, and relaxation.
  Arms: Enhanced usual care

SUMMARY:
The overarching long-term goal of the Integrative Medicine for Patient-reported Outcomes Values and Experience (IMPROVE) research program is to evaluate whether integrating a virtual mind-body programming, Integrative Medicine at Home (IM@Home), will improve patient perceived values, outcomes, and experiences as they undergo systemic cancer treatment such as chemotherapy, immunotherapy, radiotherapy, targeted agents, cytoreductive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or older
* Karnofsky score 60 or greater
* Life expectancy greater than six months
* English speaking

Additional Inclusion Criteria for Head and Neck, Thoracic, Gynecologic, Melanoma and Breast Baskets

* Patients with a diagnosis of head and neck tumors, thoracic tumors, gynecological tumors, melanoma, breast cancer, or gynecologic cancer
* Actively receiving systemic oncological treatment or radiotherapy, or within 4 weeks of radiotherapy completion or primary cytoreductive surgery
* Worst fatigue over the last 7 days rated 4 or greater on (0-10 scale)

Additional Inclusion Criteria for First Remission Gynecologic Cancer Basket

* Patients with a diagnosis or clinical suspicion of gynecologic malignancy who have completed definitive first line treatment (maintenance hormonal or targeted therapies are allowed)

Additional Inclusion Criteria for the Advanced Cancer Basket:

* Patients with a diagnosis of Stage III or IV lung cancer; any stage pancreatic cancer, unresectable cholangiocarcinoma, unresectable liver cancer, unresectable ampullary or peri-ampullary cancer, or other stage IV gastrointestinal cancer; stage III or IV ovarian or fallopian tube cancers or other stage IV gynecologic cancer; stage IV breast cancer; stage III testicular cancer or any stage IV genitourinary cancer; stage IV sarcoma; stage IV melanoma; stage IV endocrine cancer; lymphoma, myeloma, or Leukemia
* Actively receiving oncological treatment, radiotherapy or active surveillance

Additional Inclusion Criteria for the Cancer Survivor Basket:

* Completed active cancer treatment (e.g., surgery, radiation, chemotherapy) (maintenance hormonal or targeted therapies are allowed).
* Worst fatigue over the last 7 days rated 4 or greater on (0-10 scale)

Exclusion Criteria:

* Cognitive impairment that would preclude response to study assessments or require the use of Legally Authorized Representatives
* Unwilling to accept random assignment
* Concurrently enroll onto ongoing competing trials of integrative medicine interventions with symptom/toxicity as primary outcome. Note, however, patient will be allowed to enroll on other therapeutic protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Average Fatigue Severity from the Brief Fatigue Inventory (BFI) | 12 weeks
  Primary outcome will be measured by the average fatigue severity measured by the Brief Fatigue Inventory (BFI). The BFI is a 9-item instrument designed to assess one construct of fatigue severity in cancer and non-cancer populations. Three items ask patients to rate the severity of their fatigue at its "worst," "usual," and "now" during normal waking hours, with 0 being "no fatigue" and 10 being "fatigue as bad as you can imagine." Six items assess the amount that fatigue has interfered with different aspects of the patient's life during the past 24 hours. The interference items are measured on a 0-10 scale, with 0 being "does not interfere" and 10 being "completely interferes."59 A composite fatigue severity score can be found by averaging the 9 item scores.

SECONDARY OUTCOMES:
Symptom intensity as measured by Edmonton Symptom Assessment Scale (ESAS) | 12 weeks
  The ESAS is a brief self-report tool of symptom intensity, initially developed for patients with advanced cancer.61 It includes nine common symptoms of advanced cancer (pain, tiredness, nausea, depression, anxiety, drowsiness, appetite, well-being, shortness of breath), with the option of adding a tenth patient-specific symptom. It is designed to capture multidimensional symptom profiles over time by obtaining repeated quantitative measurements of symptom intensity with minimal patient burden. The original ESAS used visual analogue scales (VAS) to rate symptom intensity. A subsequent revised version replaced the VAS with 11-point numerical rating scales.
Insomnia severity as measured by Insomnia Severity Index (ISI) | 12 weeks
  The ISI has 7 items rated on a 5-point Likert response scale (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28 with higher scores representing more severe insomnia symptoms. The usual recall period is the "last month." The ISI authors suggest the following guidelines for interpreting the ISI total score: < 8, no clinically significant insomnia; 8-14, subthreshold insomnia; 15-21, clinical insomnia (moderate severity); > 21, clinical insomnia (severe). The ISI has demonstrated internal consistency, reliability, construct validity, specificity and sensitivity in a representative sample of 1670 cancer patients. The ISI has established minimally important change values to ensure that the change is not only statistically, but also clinically, meaningful to patients. A reduction of eight points has been deemed to be clinically significant improvement.
Effect of treatments on psychological distress as measured by Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  HADS is a 14-item scale with 7 items measuring depression and 7 items measuring anxiety. Each item is answered by the patient on a four-point (0-3) response category, so possible scores range from 0-21 for anxiety and depression, with higher scores indicating higher symptomatology. Established cutoffs are: 0-7 not significant; 8-10 subclinical; and 11-21 clinically significant depression/anxiety. Factor analysis showed two distinct but correlated factors of anxiety and depression. The scale scores have been shown to be both reliable and valid.
Pain as measured by Patient Reported Outcomes Measurement Information System (PROMIS®) Scale v1.2 - Global Health | 12 weeks
  Patient Reported Outcomes Measurement Information System (PROMIS®) Scale v1.2 - Global Health is a brief instrument composed of 10 items that demonstrates adequate reliability and validity as a measure of health-related QOL in general and clinical populations. Patients are asked to respond to questions 1-8 and 10 on a scale of 1-5. Question 9 is on a 0-10 scale (average pain rating). The measure yields two scores, Physical Health and Mental Health, that will be used as secondary outcomes to evaluate the effect of our interventions on QOL. These scores will be calculated using item-level calibrations based on item response theory (IRT) scaling and then transformed to T-Scores, which are standardized such that 50 represents the mean for the US general population, and the standard deviation around that mean is 10 points. Higher scores indicate better Physical and Mental Health.
Participants treatment outcome expectancy as measured by Mao Expectancy of Treatment Effects (METE) | 12 weeks
  Mao Expectancy of Treatment Effects (METE): is a four-item instrument originally developed as the Acupuncture Expectancy Scale (AES) by Mao (PI) et al. Outcome expectancy has long been considered an important predictor of treatment outcomes and has gained increasing recognition in clinical trials. It has demonstrated reliability (Cronbach's α of 0.82) and validity and is positively correlated with patient self-reported efficacy and satisfaction. The score ranges from 4 to 20, with higher scores indicating greater expectancy. We will use this measure to explore whether expectancy predicts treatment outcomes and may impact the observed differences between groups.
Satisfaction of intervention | 12 weeks
  Satisfaction will be measured through a five-point Likert scale assessing overall approval and recommendations for improvement. Trevino et al. (2020) demonstrated high engagement and satisfaction with IMS remotely delivered mind-body services, including fitness, meditation, yoga.77 Furthermore, qualitative interviews will be conducted using thematic content analysis to determine program satisfaction and triangulate quantitative data.
Recommendation of Intervention to Others | 12 weeks
  Willingness to recommend the intervention will be measured by a one-item assessment. Participants will be asked their willingness to recommend the intervention to a friend, family member, or fellow cancer patient/survivor.
Number of Treatment Disruptions | 12 weeks
  Record on treatment disruption will be extracted from MSK EMR via DataLine. This includes records on dose reduction, dose delay, and treatment discontinuation. Participants will also self-report and comment on treatment disruption in log. Dose reduction is defined as any dosage decrease or adjustment relative to dosage at the start of intended systemic regimen. Dose delay is defined as any delay or temporary stoppage in administration of systemic regimen relative to the intended schedule. Treatment discontinuation is defined as permanent discontinuation of the intended systemic regimen that does not include treatment completion during intervention. The treatment variables will be abstracted by the clinical research coordinators and adjudicated with guidance from the collaborating medical oncologists in the specific services.
Number of Unplanned medical visits | 12 weeks
  Record on unplanned medical visits to the urgent care, emergency room, and hospitalization will be patient-reported and extracted from MSK EMR via DataLine. For each unplanned medical visit, CPT code, ICD-10 code, chief complaints, and the length of stay will be collected. Unplanned medical visit data will also be tracked at partner hospitals in collaboration with ambulatory care. Participants will also self-report and comment on unplanned medical visits in log.
Participant Attendance to IM@Home Sessions | 12 weeks
  Participants will self-report attendance in a weekly log of the number and type of classes attended. Once randomized, participants will be instructed to record their attendance in the mind-body classes throughout the week. A log will be sent out through the MSK Engage, where participants can fill out their attendance at the end of each week.

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Bryl, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Bryl KL, Silverwood S, Desai K, Schobert K, Li X, Chimonas S, Mao JJ, Gillespie EF. Benefits and Challenges of a Digital Exercise and Mind-Body Program During Active Cancer Treatment: Qualitative Study of Patients' Perceptions. JMIR Cancer. 2026 Jan 16;12:e80075. doi: 10.2196/80075. PMID 41543884
- [Derived] Mao JJ, Bryl K, Gillespie EF, Green A, Hung TKW, Baser R, Panageas K, Postow MA, Daly B. Randomized clinical trial of a digital integrative medicine intervention among patients undergoing active cancer treatment. NPJ Digit Med. 2025 Jan 14;8(1):29. doi: 10.1038/s41746-024-01387-z. PMID 39809874
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org